CLINICAL TRIAL: NCT07168941
Title: Evaluation and Refinement of KF-STRIDE Into the Interview!
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Helen Genova, Associate Director, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-1238-23
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kessler Foundation STRength IDentification and Expression (KF-STRIDE) (Experimental)
  Interventions: Behavioral: KF-STRIDE
- Services as Usual (No Intervention)

INTERVENTIONS:
Behavioral: KF-STRIDE — KF Stride works to improve identification (awareness) of personal character strengths and 2) express them in a socially appropriate way during a job interview
  Arms: Kessler Foundation STRength IDentification and Expression (KF-STRIDE)

SUMMARY:
Examine the acceptability, usability, feasibility, and initial efficacy of KF-STRIDE 3.0, the data from which will serve as a basis for a future fully powered RCT

DETAILED DESCRIPTION:
Although KF-STRIDE 2.0 was designed to support youth on the spectrum, its current design may not be appropriate for adults. Thus, the current proposal will support development activities to significantly adapt KF-STRIDE 2.0 to meet the specific needs of adults with autism. As part of development, we will partner with the autism community, using mixed methodology to ensure our modifications are performed with community-engaged methods. We will invite adults with autism, family members, employers, and vocational counselors to provide feedback to guide the modifications to KF-STRIDE. We will then test the acceptability, feasibility, fidelity, and initial efficacy of KF-STRIDE 3.0 among adults on the spectrum. Obtaining employment is essential to individuals on the spectrum as it can lead to improved community integration, increased social networking, and a means to contribute to society as productive citizens. Overall, we propose to adapt a treatment that has strong potential to help adults with autism improve their job interview skills that will lead to increased employment.

ELIGIBILITY:
Inclusion Criteria:

* You live in the United States of America
* You speak English Fluently and at a 4th grade reading level

Exclusion Criteria:

* You have a history of significant psychiatric illness (like bipolar disorder, schizophrenia, or psychosis)
* You have a history of substance abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-09-10 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
20-minute long video-recorded Mock Job Interview, Autism Mock Interview Rating-Scale(A-MIRS) | Baseline, Immediate Post-Test between weeks 7 and 8
  Participants will choose 1 of 7 possible employment positions (i.e., security, childcare, culinary arts). Digital recordings will be scored by blinded raters with human resources expertise and trained to a reliable standard. Briefly, raters will rate videos using the Autism Mock Interview Rating-Scale (A-MIRS). The A-MIRS rate will rate the participant's 'likeliness to be hired' as a global rating of overall interview skill (scaled from 1= "unlikely" to 5= "very likely"). Then, raters will rate 11 interview skills (using a Likert-type scale): 1) confidence; 2) being positive; 3) professionalism; 4) showing interest; 5) honesty; 6) being hardworking; 7) working with others; 8) sharing strengths and skills; 9) sharing past experiences; 10) sharing limitations; and 11) overall rapport. A total score will be evaluated.
Work Readiness Scale | Baseline, Immediate Post-Test between weeks 7 and 8
  13 items about the perception of one's ability to work, with values ranging from 1 to 5, with higher scores meaning a better outcome.
Employment Status | Baseline, Immediate Post-Test between weeks 7 and 8
  We will examine whether the person became employed or other changes to their employment status, (employment status, hours worked, wages earned, etc.) . Yes=1, No=0

SECONDARY OUTCOMES:
World Health Organization Quality of Life abbreviated version (WHOQOL-BREF) | Baseline, Immediate Post-Test between weeks 7 and 8
  A self-report questionnaire which assesses 4 domains of quality of life (QOL): physical health, psychological health, social relationships, and environment

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No